CLINICAL TRIAL: NCT01485445
Title: An Open-label, Randomised, Replicate, Six-way Crossover, Single Dose Study to Determine the Bioequivalence of Fluticasone Furoate (FF) Inhalation Powder (Single Strip Configuration) Compared With FF Inhalation Powder (Two Strip Configuration) and Compared With FF / Vilanterol (VI) Inhalation Powder Administered Via the Novel Dry Powder Inhaler.
Brief Title: Bioequivalence Study to Compare Fluticasone Furoate (FF) 1-strip Inhaler With FF 2-strip Inhaler and With FF/Vilanterol Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 115440
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: bioequivalence; pharmacokinetics; Fluticasone Furoate; Vilanterol
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol

ARMS (3):
- Fluticasone Furoate (single strip configuration) (Experimental): 400mcg, administered as 2 inhalations of 200mcg
  Interventions: Drug: Fluticasone Furoate (200mcg unit strength)
- Fluticasone Furoate (two strip configuration) (Experimental): 400mcg, administered as 2 inhalations of 200mcg. Second strip contains lactose and magnesium stearate
  Interventions: Drug: Fluticasone Furoate (200mcg unit strength)
- Fluticasone Furoate/Vilanterol (Experimental): 400/50mcg, administered as 2 inhalations of 200/25mcg
  Interventions: Drug: Fluticasone Furoate/Vilanterol (200/25mcg unit strength)

INTERVENTIONS:
Drug: Fluticasone Furoate (200mcg unit strength) — inhalation powder
  Arms: Fluticasone Furoate (single strip configuration); Fluticasone Furoate (two strip configuration)
Drug: Fluticasone Furoate/Vilanterol (200/25mcg unit strength) — inhalation powder
  Arms: Fluticasone Furoate/Vilanterol

SUMMARY:
The purpose of this study is to determine the bioequivalence of fluticasone furoate (FF) inhalation powder (single strip configuration) compared with FF inhalation powder (two strip configuration) and compared with FF / vilanterol (VI) inhalation powder. Fluticasone furoate (FF), is being developed both as a monotherapy for the treatment of asthma and in combination with vilanterol (VI) for the treatment of asthma and Chronic Obstructive Pulmonary Disease (COPD). Thirty healthy male and female subjects will be enrolled in the study to ensure twenty-four evaluable subjects.

DETAILED DESCRIPTION:
Fluticasone furoate (FF; GW685698), a novel corticosteroid, is being developed both as a monotherapy for the treatment of asthma and in combination with vilanterol (VI; GW642444) for the treatment of asthma and COPD. The novel dry powder inhaler (NDPI) will be used to deliver both FF monotherapy and the FF/VI combination. The NDPI can be used with either a single strip or two strips, the single strip being used for FF monotherapy and two strips being used to deliver the FF/VI combination. In some previous FF monotherapy studies, including the phase IIB programme, conducted using the NDPI, the inhaler contained two strips (FF in the first strip and matched VI placebo in the second strip). This two strip configuration has been used for the majority of FF monotherapy treatment arms in previous and ongoing studies. The aim of this study is to determine the bioequivalence of FF monotherapy (single strip) compared with FF monotherapy (two strip), and to determine the bioequivalence of FF monotherapy (single strip) compared with FF/VI, administered via the NDPI. This data will facilitate the inclusion of FF monotherapy (two strip) data and FF/VI combination data to support the FF monotherapy product development. This will be a randomised, open-label, replicate, six-way crossover, single dose study in healthy male and female subjects. Thirty healthy male and female subjects will be enrolled in this study to ensure twenty-four evaluable subjects.

Pharmacokinetic samples will be taken over 36 hours. Safety will be assessed by adverse event (AE) monitoring throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 of the protocol for an appropriate period of time prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until completion of the follow-up visit.

* Body Mass Index (BMI) within the range 18.5-29.0 kg/m2 (inclusive).
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin are less than or equal to 1.5x Upper Limit of Normal (ULN) (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is less than 35%).
* Average QTcF less than 450 msec.
* Forced Expiratory Volume in 1 second (FEV1) greater than or equal to 85% predicted at screening.
* Subjects who are current non-smokers, who have not used any tobacco products in the 12 month period preceding the screening visit, and have a pack history of less than or equal to 5 pack years (number of pack years = (number of cigarettes per day/20) x number of years smoked)
* Able to satisfactorily use the novel dry powder inhaler (NDPI)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. Subjects must have signed the Informed Consent Form (ICF) prior to the commencement of any screening activities.

Exclusion Criteria:

* As a result of medical interview, physical examination or screening investigations, the principal investigator or delegate physician deems the subject unsuitable for the study. Subjects must not have a systolic blood pressure above 140 mmHg or a diastolic pressure above 90 mmHg.
* The subject has a history of breathing problems in adult life (e.g. history of asthmatic symptomatology). Screening lung function tests (FEV1) will be performed to confirm normal lung function parameters (greater than or equal to 85% predicted).
* Subjects who have suffered a lower respiratory tract infection within 4 weeks of the screening visit.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units for males or greater than 14 units for females.
* A positive pre-study drug/alcohol screen or when randomly tested during the study.
* Positive cotinine and urine alcohol test at screening or on admission to the Unit.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* The subject has taken systemic, oral or depot corticosteroids less than 12 weeks before the screening visit.
* The subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, including immediate or delayed hypersensitivity to any beta-agonist, sympathomimetic drug, or any intranasal, inhaled or systemic corticosteroid therapy; known or suspected sensitivity to the constituents of the new powder inhaler (i.e. lactose or magnesium stearate), or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates participation.
* History of severe milk protein allergy.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 30 day period.
* Pregnant females as determined by positive serum hCG test at screening or by positive serum/urine hCG test prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Vulnerable subjects (eg kept in detention) or Parexel / GSK employees

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12-21 (Actual); Primary Completion 2012-03-12 (Actual); Study Completion 2012-03-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters for Fluticasone Furoate (FF) for all study participants | 15 time points between pre-dose and 36 hours post-dose in each of the six treatment periods
  Measurement of amount of FF in the blood of study participants. From the plasma concentration-time data the following PK parameters will be determined as data permits: Area Under Curve from pre-dose to infinite time (AUC)(0-inf), Area Under Curve from pre-dose to time of last quantifiable concentration (AUC)(0-t), maximum plasma concentration (Cmax)

SECONDARY OUTCOMES:
Pharmacokinetic parameters for Fluticasone Furoate (FF) for all study participants | 15 time points between pre-dose and 36 hours post-dose in each of the six treatment periods
  Measurement of amount of FF in the blood of study participants. From the plasma concentration-time data the following PK parameters will be determined as data permits: time to maximum plasma concentration (tmax), half-life (t1/2)
Adverse events (AEs) for all study participants | From the start of first dosing until follow-up (approximately 7 weeks per subject)
  Measurement of types of AEs reported, severity and relationship to study drug

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115440 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115440?search=study&search_terms=115440#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115440 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register